CLINICAL TRIAL: NCT07189754
Title: A Randomized, Double-Blind Placebo Controlled Study to Assess the Effects of an Oroxylum Indicum Extract (Sabroxy™) on Cognitive Function in Adults With Self-reported, Mild Cognitive Impairmentx
Brief Title: A Study of Sabroxy™ (Oroxylum Indicum Extract) for Improving Cognitive Function in Adults With Mild Memory Concerns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTC2020-002
Record Dates: First submitted 2025-09-11; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment (MCI); Cognitive Dysfunction, Cognitive Disorder; Memory Problems
Keywords: Computerized Cognitive Test (COMPASS); Montreal Cognitive Assessment (MoCA); Oroxylum indicum; Cognitive Performance; Sabroxy™; Cognitive Function; Brain-Derived Neurotrophic Factor (BDNF); Memory; Attention
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sabroxy™ (Oroxylum indicum extract) (Active Comparator): Consume one capsule twice daily, after a meal.
  Interventions: Dietary Supplement: Sabroxy™ (Oroxylum indicum extract)
- Placebo (Inactive capsule) (Placebo Comparator): Consume one capsule twice daily, after a meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sabroxy™ (Oroxylum indicum extract) — Sabroxy™ is a standardized extract derived from the bark of Oroxylum indicum. In this study, participants will receive Sabroxy™ in capsule form. Each capsule contains a fixed dose of the extract and will be administered orally at a regimen of one capsule twice daily after meals for 12 weeks. The supplement is provided in visually identical containers to maintain blinding and is compared to a placebo control. The intervention is designed to evaluate potential improvements in cognitive function, including memory, attention, and executive performance, as well as effects on circulating Brain-Derived Neurotrophic Factor (BDNF) levels.
  Other Names: Oroxylum indicum extract; Sabroxy™
  Arms: Sabroxy™ (Oroxylum indicum extract)
Other: Placebo — The placebo is an inert capsule formulated to be visually identical to the Sabroxy™ capsules in size, shape, color, and packaging. It contains inactive ingredients only, with no active botanical extract. The placebo will be administered orally at the same regimen as the active intervention: one capsule taken twice daily after meals for 12 weeks. The use of a placebo ensures blinding of participants and study staff, allowing accurate comparison of cognitive and biomarker outcomes between groups.
  Other Names: Inactive capsule; Look-alike capsule
  Arms: Placebo (Inactive capsule)

SUMMARY:
This study is testing whether Sabroxy™ (Oroxylum indicum extract) can improve memory and thinking in older adults who report mild problems with their cognition. The study will also measure levels of a protein in the blood called BDNF (Brain-Derived Neurotrophic Factor), which is linked to brain health.

The main questions are:

Does taking Sabroxy™ improve memory, focus, and overall cognitive performance compared to placebo (a capsule that looks the same but has no active ingredient)?

Does Sabroxy™ increase levels of BDNF in the blood?

About 80 participants between the ages of 60 and 85 will take part. All participants will be randomly assigned to receive either Sabroxy™ or placebo twice daily for 12 weeks. Neither the participants nor the researchers will know which group they are in (double-blind design).

During the study, participants will:

Take one capsule twice daily after meals.

Complete computerized cognitive tests (COMPASS), interviews with the Montreal Cognitive Assessment (MoCA), and self-assessment questionnaires on memory and thinking.

Provide blood samples to measure BDNF.

Attend 4 clinic visits (baseline, week 4, week 8, and week 12).

Keep a daily diary to track product use and study compliance.

The goal is to see whether Sabroxy™ can safely and effectively support cognitive health in older adults with mild memory concerns.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effects of Sabroxy™ (Oroxylum indicum extract) on cognitive function in adults with self-reported, mild cognitive impairment.

Approximately 84 participants will be recruited, with a goal of 80 completing the study. Participants will be between 60-85 years old, in generally good health, and living independently. Eligible participants must report concerns about their memory or thinking, confirmed with a screening test (MoCA).

After screening and baseline assessments, participants will be randomly assigned to receive either Sabroxy™ or placebo. Both products will look identical to ensure blinding. Participants will take one capsule twice daily, after meals, for 12 weeks.

The study assessments include:

Computerized Mental Performance Assessment (COMPASS): tests of memory, attention, and reaction time.

Montreal Cognitive Assessment (MoCA): an interviewer-administered cognitive test.

Mild Cognitive Impairment Questionnaire: a self-reported measure of memory and thinking concerns.

Blood samples: to measure Brain-Derived Neurotrophic Factor (BDNF) at baseline and week 12.

Daily diaries and capsule counts: to monitor adherence.

The visit schedule is as follows:

Baseline (Visit 1): Screening, informed consent, eligibility check, cognitive testing, blood draw, product distribution, and diary instructions.

Week 4 (Visit 2): Product count, diary review, questionnaire.

Week 8 (Visit 3): Product count, diary review, questionnaire.

Week 12 (Visit 4): Cognitive testing, blood draw, questionnaire, product return, diary review.

Statistical analyses will compare changes in cognitive performance and BDNF levels between the Sabroxy™ and placebo groups.

This study will provide important information about the potential of Sabroxy™ to support memory and brain health in older adults with mild cognitive concerns.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male and female), 60 to 85 years old

Residing in independent living accommodation

Subjective reports of memory or cognitive impairment (answering "yes" to at least one of the following):

Do you feel your memory and thinking is getting worse?

Do you feel your memory and thinking has become worse over the past 2-3 years?

Are you concerned about your decline in memory and thinking?

Modified Montreal Cognitive Assessment (MoCA) score consistent with mild impairment

Non-smoker

Body Mass Index (BMI) between 18 and 35 kg/m²

No plans to commence new treatments over the study period

Understands and is willing to comply with study procedures

Provides signed and dated informed consent

Exclusion Criteria:

* Diagnosis of dementia (per NIA/AA criteria)

Uncontrolled hypertension, cardiovascular disease (MI, angina, CHF), bleeding disorders, type I diabetes, glaucoma, renal/hepatic disease, pulmonary or significant GI disease, gallbladder/biliary disease, or neurodegenerative/neurological disease

Significant psychiatric disorder (schizophrenia, bipolar disorder, OCD, personality disorder)

History of stroke, seizures, or head injury with loss of consciousness

Moderate-to-severe depression or anxiety (per Depression, Anxiety, Stress Scale)

Regular use of anticoagulants, anticholinergics, acetylcholinesterase inhibitors, or steroids

Medication change in past 3 months or expected changes during study

Use of vitamins or herbal supplements that may affect cognition

Current or recent (12 months) illicit drug abuse

Alcohol intake >14 drinks/week

Significant surgery in the last year

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) total score | Baseline and Week 12
  The Montreal Cognitive Assessment (MoCA) is a 30-point interviewer-administered test assessing memory, attention, visuospatial ability, language, and executive function. Scores range from 0 to 30, with higher scores indicating better cognitive function (a score ≥26 is generally considered normal). The mean change from baseline to Week 12 will be compared between the Sabroxy™ and placebo groups.
Change in COMPASS accuracy composite (percent correct) | Baseline and Week 12
  The Computerized Mental Performance Assessment System (COMPASS) provides accuracy scores (% correct) across cognitive subtests (e.g., memory recognition, working memory). Composite accuracy is reported as the mean percentage correct across prespecified subtests. Scores range from 0% to 100%, with higher percentages indicating better accuracy/performance. The mean change from baseline to Week 12 will be compared between the Sabroxy™ and placebo groups.
Change in COMPASS mean reaction time (milliseconds) | Baseline and Week 12
  The Computerized Mental Performance Assessment System (COMPASS) measures reaction time in milliseconds (ms) across attention and response tasks. Reaction time is a continuous measure (theoretical range: 0 ms to no fixed upper limit). Lower values indicate faster and therefore better performance. Results will be reported as mean milliseconds and mean change from baseline.

SECONDARY OUTCOMES:
Change in Mild Cognitive Impairment Questionnaire (self-reported cognitive function) total score | Baseline, Week 4, Week 8, Week 12
  The Mild Cognitive Impairment Questionnaire is a self-report tool where participants rate memory and thinking difficulties over the past 4 weeks. Responses are recorded on a 5-point Likert scale (1 = Never, 5 = Always) across multiple items. Scores are summed to generate a total score, with the minimum possible score = [lowest possible total, e.g., number of items × 1] and maximum = [number of items × 5]. Higher scores indicate worse self-reported cognitive function (greater impairment). Mean change from baseline to Weeks 4, 8, and 12 will be compared between Sabroxy™ and placebo groups.
Change in Brain-Derived Neurotrophic Factor (BDNF) Levels | Baseline and Week 12
  Blood samples will be collected to measure serum BDNF levels. Mean change from baseline to Week 12 will be compared between Sabroxy™ and placebo groups.
Compliance with investigational product by capsule count | Week 4, Week 8, Week 12
  Compliance will be assessed by counting returned capsules at each visit. Compliance percentage will be calculated as:
  (number of capsules actually taken ÷ number of capsules expected to be taken) × 100(number of capsules actually taken ÷ number of capsules expected to be taken) × 100(number of capsules actually taken ÷ number of capsules expected to be taken)×100. The mean compliance percentage will be compared across groups. Unit of Measure: Percent (%)
Incidence of Treatment-Emergent Adverse Events (AEs) | Baseline through Week 12
  Safety will be assessed by recording all treatment-emergent adverse events reported or observed from baseline through Week 12. Results will be reported as the number and percentage of participants experiencing at least one AE.
Compliance with investigational product by daily diary review | Week 4, Week 8, Week 12
  Compliance will also be assessed by reviewing participant daily diaries documenting capsule intake. Compliance percentage will be calculated as:
  (number of days capsule intake recorded ÷ number of days expected)×100(number of days capsule intake recorded ÷ number of days expected) × 100(number of days capsule intake recorded ÷ number of days expected)×100.
  The mean compliance percentage will be compared across groups. Unit of Measure: Percent (%)
Incidence of Serious Adverse Events (SAEs) | Baseline through Week 12
  Serious adverse events will be recorded throughout the study. Results will be reported as the number and percentage of participants experiencing at least one SAE. Unit of Measure: Number of participants.
Incidence of Participant-Reported Side Effects | Baseline through Week 12
  Tolerability will be assessed through participant-reported side effects, captured via direct questioning and diary review. Results will be reported as the number and percentage of participants reporting at least one side effect. Unit of Measure: Number of participants.
Number of Discontinuations Due to Adverse Events | Baseline through Week 12
  The number of participants who discontinue the study due to adverse events will be recorded and compared between treatment groups.
  Unit of Measure: Number of participants

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No